CLINICAL TRIAL: NCT02443103
Title: Exploratory Pilot Study Evaluating the Biologic Activity of Guanabenz in Bone Metastasis
Brief Title: Study Evaluating the Biologic Activity of Guanabenz in Bone Metastasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Kathy Miller (Other)
Responsible Party: Sponsor-Investigator, Kathy Miller, Full Professor of Medicine and Sheila D. Ward Scholar, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0506
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Bone Cancer; Metastasis
Keywords: pilot study; guanabenz acetate
MeSH Terms: conditions — Bone Neoplasms; Neoplasm Metastasis | interventions — Guanabenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Guanabenz (Experimental)
  Interventions: Drug: Guanabenz acetate

INTERVENTIONS:
Drug: Guanabenz acetate

SUMMARY:
This study will explore the biologic activity of guanabenz in reducing bone turn over in solid tumor patients with bone metastasis. If successful, this repurposing of an already, generic drug could benefit patients faster than manufacturing a novel expensive compound.

DETAILED DESCRIPTION:
OBJECTIVES Primary Objective: Evaluate the biologic effect of guanabenz on markers of bone formation and bone resorption in patients with solid tumors and bone metastasis.

Secondary Objectives: (1) Compare guanabenz exposure in patients based on limited PK sampling to activity observed in previous pre-clinical studies; (2) Assess the safety/tolerability of guanabenz; and (3) Evaluate the biologic effect of guanabenz on bone metabolism markers.

Tertiary Objective: Compare change in bone turn over markers (formation, resorption and metabolism) achieved with guanabenz to change in bone turn over markers with standard of care (bisphosphonate/denosumab).

STUDY DESIGN This is an exploratory pilot study evaluating the biologic effect of guanabenz bone formation and bone resorption markers in patients with solid tumors and bone metastasis.

PROCEDURES All registered patients will receive oral guanabenz the first two months prior to the start of any standard of care skeletal protective therapy. All patients on study will receive standard of care systemic treatment for their underlying solid malignancy as deemed necessary by their treating physician. Guanabenz will be administered concurrently with any primary cancer systemic treatment. However patients will withhold standard of care bone directed therapy for 8 weeks. The study will exclude patients in immediate need of such treatment. Patients experiencing skeletal related events while on study will be withdrawn. Delaying standard of care skeletal therapy for 2 months will not be considered a major deviation as long as such therapy is delayed for a necessary purpose as deemed by the treating physician.

Patients with known hypertension and on antihypertensive medications at study enrollment will be eligible to participate. Antihypertensive medications will not be changed as a result of study enrollment unless deemed necessary by the treating physician; only the dose of guanabenz will be adjusted.

TREATMENT Patients will begin taking 8 mg by mouth (PO) at bed time (HS) starting day 1 for one week. The dose will be increased to 8 mg PO twice a day (BID) (8 mg daily morning (QAM) and 8 mg daily evening (QPM) for a total of 16 mg) on day 8 (+/-3 days), then increased to 8 mg PO QAM 16 mg PO QPM (total of 24 mg) on day 15 (+/- 3 days), then increased to 16 mg PO BID (16 mg QAM and 16 mg QPM for a total of 32 mg) on day 22. Patients will continue on their maximum tolerated dose (MTD) until day 56 (+/- 3 days). The dose will be weaned for patients receiving more than 8 mg daily after completing week 8 when the standard of care skeletal protective therapy begins. Guanabenz will be weaned off by week 11, and patients will continue standard of care skeletal protective therapy as deemed necessary by the treating physician.

To ensure patient safety during dose escalation and throughout the study, patients will be provided and taught the use of home blood pressure (BP) monitoring. We will instruct patients to check their BP 2 hours after each guanabenz dose escalation and at least three times weekly. Patients will maintain a diary of BP results during the dose escalation phase. Patients will report any hypotensive measurement to their research nurse defined as at least two readings less than < 100/60 mm Hg in sitting position taken more than 30 min apart.

At each visit, blood pressure and adverse events will be assessed. Dose escalation will continue with guanabenz if BP >= 110/70 mm Hg and/or until unacceptable toxicity.

Guanabenz should be taken as instructed on an empty stomach. If the patient misses a dose of guanabenz, he/she can take the missing dose no later than 3 hours after instructed time and then continue as scheduled.

On day 57 (+/- 3 days), all study patients start the guanabenz wean. All patients will receive ongoing standard of care skeletal protective therapy (denosumab/zometa) as determined by the treating physician at the beginning of the weaning phase.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Solid organ malignancy with documented bone metastasis by imaging
4. Adequate liver function (serum total bilirubin <= 3 and AST/ALT <= 3 times the upper normal limit)
5. Adequate renal function (serum creatinine <= 2mg/dL)
6. Ability to swallow oral tablets
7. Females of childbearing potential must have a negative pregnancy test <= 28 days prior to registration. All females of childbearing potential who are sexually active, must agree to use a highly reliable method of contraception to prevent pregnancy. These include abstinence, partner with previous vasectomy, placement of an intrauterine device (IUD), condom with spermicidal foam/gel/film/cream/suppository, diaphragm or cervical vault cap, or hormonal birth control (pills or injections).

   NOTE: Females are considered of childbearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal (> 12 months since last menses).
8. Patients are permitted to participate in other clinical trials while participating in this trial.
9. Patients will receive standard of care systemic treatment for underlying solid malignancy as deemed necessary by treating physician.

Exclusion Criteria:

1. No prior history of bisphosphonate ordenosumab use in the past 12 months
2. No history of SRE within past 3 months

   1. Excruciating bone pain requiring RT
   2. Cord compression
   3. Hypercalcemia [serum calcium >10.5]
   4. Pathologic fracture
3. No history of Paget's disease
4. No history of epilepsy/seizures
5. No history of hypotension (defined as resting systolic blood pressure of < 110 mm Hg or diastolic blood pressure of < 70 mm Hg) or orthostasis (defined as drop in systolic blood pressure of >20 mm Hg or increase in HR of > 20 from supine to standing position).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University (IU) School of Medicine, Department of Medicine; IU Health
Locations (4):
- United States (4):
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney & Lois Eskenazi Hospital, Indianapolis, Indiana
  - Spring Mill Medical Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on enrolling 15 patients. Due to poor accrual and the decision that the approach with this agent is not feasible, the study was closed with 4 patients enrolled.
Groups:
- Guanabenz: Guanabenz (titrate up from 8mg PO QPM to 16mg PO BID max dose)
Period: Overall Study
Arm/Group | Guanabenz
Started | 4
Completed | 1
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Guanabenz
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (2.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Bone Turnover Markers-bone Formation and Bone Resorption
Description: Number of patients who had blood specimens taken to collect and evaluate markers of bone formation and bone resorption. Note - due to poor accrual and early closure, bone marker data was not collected.
Time Frame: Day 0, Week 8, Week 12
Population: All patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit with bone marker information available.
Arm/Group | Guanabenz
Number analyzed (Participants) | 0

2. Secondary Outcome: Treatment Related Adverse Events
Description: Number of unique patients who had a treatment related (possible, probable or definite) adverse events.
Time Frame: Up to 1 year
Population: All patients enrolled and received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Guanabenz
Number analyzed (Participants) | 4
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Guanabenz
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guanabenz (N=4)
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Dizziness (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Hot flashes (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to poor accrual and the early closure, results were not obtained for the bone marker and pharmacokinetics analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes